CLINICAL TRIAL: NCT07275151
Title: Repeatable Evaluation of Functional Intra-procedural Signals for Effect in Pulsed Field Ablation. REFINE-PFA
Brief Title: Repeatable Evaluation of Functional Intra-procedural Signals for Effect in Pulsed Field Ablation REFINE-PFA
Acronym: REFINE-PFA
Status: Not yet recruiting | Type: Observational
Sponsor: CathVision ApS (Industry)
Responsible Party: Sponsor
Other Study IDs: CVPFA-002
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Pulmonary vein isolation ablation — Electrical isolation of the pulmonary veins to treat atrial fibrillation

SUMMARY:
The study is a prospective, exploratory observational study with the ECGenius® System and the PFAnalyzer software module in PFA cases using the FaraPulse PFA system. The cohort will be patients with paroxysmal or persistent atrial fibrillation (AF) who undergo PVI using this system.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common cardiac arrhythmia and is associated with a five-fold increase in stroke. Pulmonary vein isolation (PVI) has become accepted treatment for AF. Historically, this has been achieved using thermal energy. However, more recently a new energy source known as pulsed field ablation (PFA) has been introduced. As PFA is tissue selective, it preserves the function of nearby structures such as the esophagus and phrenic nerve making it safer to use. As PFA is delivered in short bursts of high energy, it is also more efficient and leads to shorter procedures. However, the catheters designed to deliver PFA differ to those used previously and may not provide the same information about efficacy, making it more difficult for the operator to ascertain if the lesions have durably isolated the pulmonary vein. This exploratory observational study will assess the utility of a software module designed to measure the local potential derived from the unipolar electrogram recorded at the electrode that has delivered the PFA. During the procedure, the study will collect data only and all analysis of the output of the PFAnalyzer software module will be made off-line once the procedure is complete. The operator will follow the hospital's standard of care during the procedure, and the software module will not be used to guide therapy, nor will there be any additional time added to the procedure.

The study is a prospective, exploratory observational study with the ECGenius® System and the PFAnalyzer software module in PFA cases using the FaraPulse PFA system. The cohort will be patients with paroxysmal or persistent atrial fibrillation (AF) who undergo PVI using this system.

ELIGIBILITY:
Inclusion Criteria:

Eligible subjects will meet all of the following inclusion criteria:

1. Subjects undergoing first time pulmonary vein isolation indicated by investigator for the treatment of atrial fibrillation.
2. Male or non-pregnant female aged ≥21 years.
3. Able and willing to provide written informed consent prior to any clinical investigation related procedure.
4. Subjects in sinus rhythm at the time of the PFA application.

Exclusion Criteria:

Eligible subjects will not meet any of the following exclusion criteria:

1. Pregnant or nursing subjects.
2. Current participation in another investigational drug or device study that interferes with this study.
3. Subjects who, in the opinion of the investigator, are not candidates for this study.
4. Patients who have had a prior ablation procedure.
5. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.
6. Life expectancy is less than 12 months, in the opinion of the investigator.
7. Subjects who, in the opinion of the investigator, are considered part of any vulnerable population.
8. Subjects unlikely to be in sinus rhythm at the time of the procedure or unlikely to remain in sinus rhythm after cardioversion

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with paroxysmal atrial fibrillation and referred for a denovo pulmonary vein isolation ablation procedure using pulsed field ablation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pulmonary vein isolation | intra-procedural
  assess the agreement between pulmonary vein isolation status as determined by the operator using entrance block as well as exit block during PV pacing and as classified by the PFAnalyzer software based on unipolar local potential characteristics analyzed off-line, post procedure.

SECONDARY OUTCOMES:
Clinical utility | intra-procedural
  Assessment of the operators' subjective experience of clinical utility of the PFAnalyzer software measured through a 17-item questionnaire.
Identify a clinically meaningful threshold for residual potentials after PFA delivery. | intra-procedural
  Identify a clinically meaningful threshold for residual potentials after PFA delivery by comparing the amplitude of manually expert labelled local potentials to none local potential signals.
Feasibility of guiding rotation | intra-procedural
  Determine the feasibility of using PFAnalyzer to assist in optimizing rotation and placement of the catheter by measuring changes in local potential amplitude during rotation.

CONTACTS AND LOCATIONS:
Overall Officials: Suneet Mittal, MD, Principal Investigator — Valley Health Systems

IPD SHARING:
Plan to Share IPD: No